CLINICAL TRIAL: NCT00060684
Title: A Phase I Trial of BBR 2778 in Combination With Fludarabine, Dexamethasone and Rituximab in the Treatment of Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Dose Ranging Trial for Pixantrone in the FND-R Variant Regimen in Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Gabriella Camboni, M.D., Cell Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA I-06; NCT00057772 (obsolete NCT alias)
Record Dates: First submitted 2003-05-09; First posted 2003-05-12 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2008-09

CONDITIONS: Lymphoma, Low-Grade; Lymphoma, Small Lymphocytic; Lymphoma, Mixed-Cell, Follicular; Lymphoma, Small Cleaved-Cell, Follicular
Keywords: Pixantrone; BBR 2778; chemotherapy; DNA Intercalator; mitoxantrone; fludarabine; dexamethasone; Rituximab; Rituxan; Mabthera; monoclonal antibody; antibody; NHL; Non-Hodgkin's lymphoma; indolent; low grade; Novuspharma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — pixantrone; fludarabine; Dexamethasone; Rituximab

INTERVENTIONS:
Drug: Pixantrone (BBR 2778)
Drug: fludarabine
Drug: dexamethasone
Drug: rituximab

SUMMARY:
The aim of this trial is to determine the appropriate dose of pixantrone to be used in this combination and obtain data on the combination's safety and activity profile.

DETAILED DESCRIPTION:
The FND-R regimen is commonly used in the treatment of indolent Non-Hodgkin's lymphoma (NHL) and contains the chemotherapy agents mitoxantrone, fludarabine, dexamethasone (a steroid) and the monoclonal antibody rituximab. In this trial we are replacing mitoxantrone with pixantrone, an agent with a similar chemical structure (both agents are DNA intercalators). The trial is being run in patients with relapsed or refractory indolent NHL and aims to define the appropriate dose of pixantrone to be used in this combination, as well as to obtain data on pixantrone's safety and activity profile in combination with these drugs.

This trial is expected to recruit up to 30 patients in the USA. Patients will be treated with the drug combination for up to eight months and then followed closely in the four-week period after the last administration. After that, patients will receive physician check-ups every three months.

ELIGIBILITY:
Inclusion criteria

* Patients with relapsed or refractory indolent (low-grade) NHL
* Who have received 1-3 prior treatments with chemotherapy

Exclusion criteria

* Patients previously treated with fludarabine
* Prior treatment with rituximab (Rituxan), unless there was a complete response (CR) or partial response (PR) to that treatment
* Patients known to have an allergic reaction to rituximab, or to murine proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-12; Primary Completion 2005-01 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Determine MTD | Per cycle

SECONDARY OUTCOMES:
Establish safety profile | per cycle

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stromatt, MD, Study Director — CTI BioPharma
Locations (4):
- United States (4):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - New Mexico Onc/Hem Consultants, Inc., Albuquerque, New Mexico
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Srokowski TP, Liebmann JE, Modiano MR, Cohen GI, Pro B, Romaguera JE, Kuepfer C, Singer JW, Fayad LE. Pixantrone dimaleate in combination with fludarabine, dexamethasone, and rituximab in patients with relapsed or refractory indolent non-Hodgkin lymphoma: phase 1 study with a dose-expansion cohort. Cancer. 2011 Nov 15;117(22):5067-73. doi: 10.1002/cncr.26121. Epub 2011 Jun 16. PMID 21681734